CLINICAL TRIAL: NCT02210104
Title: Phase I Study of Cellular Adoptive Immunotherapy Using Autologous CD4+ NY-ESO-1-Specific T Cells and Anti-CTLA4 For Patients With NY-ESO-1-Expressing Tumors
Brief Title: Adoptive Therapy Using Antigen-Specific CD4 T-Cells
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Issues with tetramer staining
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0669; R01CA104711-09 (NIH)
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Melanoma; Sarcoma
Keywords: Melanoma; Sarcoma; Mixed round cell liposarcoma; Advanced; Metastatic; Immunotherapy; Ipilimumab; Yervoy; BMS-734016; MDX010; Cyclophosphamide; Cytoxan; Neosar; CD4+T Cells
MeSH Terms: conditions — Melanoma; Sarcoma; Neoplasm Metastasis | interventions — Ipilimumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ipilimumab + Cyclophosphamide + CD4+T Cells (Experimental): Starting Dose of Ipilimumab 1.0 mg /kg by vein on Days 1, 22, 43, and 64. Cyclophosphamide 300 mg/m2 administered intravenously 2 days prior to T cell infusion as an outpatient procedure. Antigen-specific CD4+ T cells administered at a dose 10^10 cells/m^2.
  Interventions: Drug: Ipilimumab; Drug: Cyclophosphamide; Biological: CD4+ T cells

INTERVENTIONS:
Drug: Ipilimumab — Starting Dose of Ipilimumab: 1.0 mg /kg by vein on Days 1, 22, 43, and 64.
  Other Names: Yervoy; BMS-734016; MDX010
Drug: Cyclophosphamide — 300 mg/m2 administered intravenously 2 days prior to T cell infusion.
  Other Names: Cytoxan; Neosar
Biological: CD4+ T cells — Antigen-specific CD4+ T cells administered at a dose of 10^10 cells/m^2 on Day 0.

SUMMARY:
The goal of this clinical research study is to learn about the safety of giving CD4+T cells with ipilimumab and cyclophosphamide.

CD4+T cells are a type of white blood cell. Researchers grow the T cells in the laboratory, and they are designed to find cancer cells and may kill them.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. The first 3 or 6 participants will receive a lower dose of ipilimumab. If there are no intolerable side effects, then the second group of 6 participants will receive a higher dose of ipilimumab.

All study participants will receive the same dose level of cyclophosphamide and the CD4+T cells.

Study Drug Administration:

You will receive cyclophosphamide by vein over about 30-60 minutes on Day -2 (2 days before you receive the CD4+T cells). If the doctor thinks it is needed, you will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

On Day 0, you will receive the CD4+T cells by vein over about 30-60 minutes. You will stay in the hospital overnight after the dose.

On Days 1, 22, 43, and 64, you will receive ipilimumab by vein over about 90 minutes.

Study Visits:

Within 2-4 weeks before you receive the CD4+T cells:

* You will have a physical exam.
* Blood (about 5½ tablespoons) will be drawn for routine tests, immune system tests, and tests on how long the T-cells survive in your body.
* You will have a computed tomography (CT) scan or x-rays to check the status of the disease.

On Day -2:

* You will have a physical exam.
* Blood (about 1 tablespoon) will be drawn for routine tests. This routine blood draw will include a pregnancy test if you can become pregnant.

On Day 1:

* You will have a physical exam.
* Blood (about 1 tablespoon) will be drawn for routine tests.

On Days 0, 7, 14, 22, 28, 35, 43, 49, and 56:

* You will have a physical exam.
* Blood (about 5½ tablespoons) will be drawn for routine tests, immune system tests, and tests on how long the T-cells survive in your body.

On Day 3, blood (about 5½ tablespoons) will be drawn for routine tests, immune system tests, and tests on how long the T-cells survive in your body.

Between Day 35 and 42 and again between Day 77 and 84, you will have a CT scan or x-rays to check the status of the disease.

The study tests may be repeated or you may have additional tests performed anytime the doctor thinks it is needed.

Some of the study tests may be done at your local clinic if you cannot return to MD Anderson. The study staff will discuss this with you.

Length of Study Drug Dosing:

Your last study drug dose will be on Day 64. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up.

End-of-Study-Drug-Dosing Visit:

On Day 64:

* You will have a physical exam.
* Blood (about 5½ tablespoons) will be drawn for routine tests, immune system tests, and tests on how long the T-cells survive in your body.

Follow-Up:

On Days 70, 77, 84, 105, 126, 147, and 168:

* You will have a physical exam.
* Blood (about 5½ tablespoons) will be drawn for routine tests, immune system tests, and tests on how long the T-cells survive in your body.

Every 3 months after Day 84, unless the disease gets worse or you start another cancer therapy, you will have a CT scan or x-rays to check the status of the disease. Every 3 months for up to 5 years, the study staff will call you or ask your doctor how you are doing. If you are called, the calls should last about 10-15 minutes.

If the doctor thinks it is needed to confirm the status of the disease, blood (about 1½ tablespoons) will be drawn every 3 months for up to 1 year.

If the doctor thinks it is needed, you will return to the clinic every 4-6 weeks starting after Day 168 or as often as the doctor thinks is needed. These visits will stop if the T-cells disappear or if the disease gets worse. Blood (about 5½ tablespoons) will be drawn for routine tests, immune system tests, and tests on how long the T-cells survive in your body.

This is an investigational study. CD4+T cells are not FDA approved or commercially available. They are currently being used for research purposes only. Cyclophosphamide is FDA approved and commercially available for the way it is being used in this study. Ipilimumab is FDA approved and commercially available for the treatment of melanoma, but not for sarcoma. The study doctor can explain how the study drugs are designed to work.

Up to 12 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologic documentation of melanoma, synovial sarcoma or mixed round cell liposarcoma concurrent with the diagnosis of metastatic disease.
2. Tumor expression of NY-ESO-1 (2+ staining or > 25%) by IHC.
3. Male or female subjects ≥18 years of age.
4. Expression of HLA-DPB1*0401
5. Eastern Cooperative Oncology Group (ECOG)/ Zubrod performance status of '0-1' .
6. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized. Suggested precautions should be used to minimize the risk or pregnancy for at least 1 month before start of therapy, and while women are on study for up to 3 months after T cell infusion, and at least 8 weeks after the study drug is stopped. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal
7. Men must be willing and able to use an acceptable method of birth control, for at least 3 months after completion of the study, if their sexual partners are WOCBP.
8. Willing and able to give informed consent.
9. Adequate venous access - consider peripherally inserted central venous catheter (PICC) or central line
10. Bi-dimensionally measurable disease by palpation on clinical exam, or radiographic imaging (X-ray or CT scan)
11. At least 4 weeks must have elapsed since the last chemotherapy, immunotherapy, radiotherapy, or major surgery.
12. At least 6 weeks must have elapsed since the last nitrosoureas, mitomycin C and liposomal doxorubicin
13. Toxicity related to prior therapy must either have returned to < or equal to grade 1, baseline, or been deemed irreversible

Exclusion Criteria:

1. Patients with active infections or oral temperature > 38.2 C within 71 hours of Leukapheresis. The procedure may be deferred.
2. Patients with Hct <30%, white blood count (WBC) <2500/uL and platelets <50,000 immediately prior to Leukapheresis. The procedure may be deferred.
3. Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix.
4. Complete blood count (CBC) and Chemistry profile prior to cyclophosphamide and T cell infusions: WBC < 2000/uL Hct < 24% or Hb < 8 g/dL absolute neutrophil count (ANC) < 1000 Platelets < 50,000 Creatinine > 3.0 x ULN AST/ALT > 2.5 x ULN Bilirubin > 3 x ULN
5. Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception. Women of childbearing potential with a positive pregnancy test within 3 days prior to entry.
6. Clinically significant pulmonary dysfunction, as determined by medical history and physical exam. Patients so identified will undergo pulmonary functions testing and those with FEV1 < 2.0 L or DLco (corr for Hgb) < 75% will be excluded.
7. Significant cardiovascular abnormalities as defined by any one of the following: Congestive heart failure, Clinically significant hypotension, Symptoms of coronary artery disease, Presence of cardiac arrhythmias on EKG requiring drug therapy,Ejection fraction < 50 % (echocardiogram or MUGA).
8. Active and untreated central nervous system (CNS) metastasis (including metastasis identified during screening MRI or contrast CT).
9. Autoimmune disease: Patients with a history of Inflammatory Bowel Disease are excluded from this study, as are patients with a history of autoimmune disease (e.g. Systemic Lupus Erythematosus, vasculitis, infiltrating lung disease) whose possible progression during treatment would be considered by the Investigator to be unacceptable.
10. Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea.
11. Positive screening tests for HIV, Hep B, and Hep C. If positive results are not indicative of true active or chronic infection, the patient can be treated.
12. Steroids are not permitted 3 days prior to T cell infusion and concurrently during therapy.
13. Any non-oncology vaccine therapy used for the prevention of infectious disease within 1 month before or after any ipilimumab dose.
14. No prisoners or children will be enrolled on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Adoptively Transferred CD4 T Cells | 12 weeks after T cell infusion
  (MTD) defined as dose level below that at which excessive toxicity was observed. Dose limiting toxicity: Any ≥ Grade 2 eye pain or reduction of visual acuity that does not respond to topical therapy and does not improve to ≤ Grade 1 severity within 2 weeks of starting therapy requires systemic treatment; Any ≥ Grade 3 bronchospasm or other hypersensitivity reaction; Any adverse event, laboratory abnormality or intercurrent illness which, in the judgment of the Investigator, presents a substantial clinical risk to the patient with continued dosing; Any other ≥ Grade 3 non-skin related adverse event.

SECONDARY OUTCOMES:
Clinical Response | 6 weeks after T cell infusion
  Complete response (CR) defined as total regression of all tumors, a partial response (PR) as 30% or greater decrease in the sum of the longest diameter of target lesions and progressive disease (PD) as 20% increase in the sum of the longest diameter of target lesions (modified world health organization criteria or mWHO. Radiographic imaging (as clinically indicated) and clinical assessment of residual disease compared with pre-infusion assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Cassian Yee, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org